# Diabetic Retinopathy Clinical Research Network (DRCR.net)

# PROMINENT-Eye Ancillary Study: Diabetic Retinopathy Outcomes in a Randomized Trial of Pemafibrate Versus Placebo

Protocol Amendment 1 Version 2.0

March 14, 2018

# **Signature Page**

| JCHR Principal Investigator |
|-------------------------------------------------|
| Name, degree |
| Signature / Date |
| External Sponsor |
| (Kowa Research Institute, Inc.) |
| Name, degree |
| Signature / Date |
| Center for Cardiovascular Disease<br>Prevention |
| Name, degree |
| Signature / Date |

# **Table of Contents**

| Abbreviations | 5 |
|---|---|
| INTRODUCTION 1.1 Diabatic Patinopathy Complications and Dublic Health Impact | 6 |
| 1.1 Diabetic Retinopathy Complications and Public Health Impact | 6 |
| 1.2 Preventing DR Onset and Worsening | |
| 1.3 Limitations of Current Treatments for PDR and DME | |
| 1.4 Rationale for PPARα Therapy for DR Worsening | |
| 1.5 Pemafibrate and the Ongoing PROMINENT trial | |
| 1.6 Summary of Protocol Rationale | |
| 1.7 Study Objective | |
| 1.8 Study Design and Synopsis of Protocol | |
| 1.9 General Considerations | |
| STUDY PARTICIPANT ELIGIBILITY AND ENROLLMENT | 14 |
| 2.1 Identifying Eligible Participants and Obtaining Informed Consent | 14 |
| 2.2 Subject Eligibility and Exclusion Criteria | |
| 2.2.1 Eligibility Criteria | |
| 2.2.2 Study Eye Criteria: | |
| 2.3 Screening Evaluation and Baseline Testing | |
| 2.3.1 Ocular Historical Information | |
| 2.3.2 Baseline Testing Procedures | |
| FOLLOW-UP VISITS | |
| 3.1 Visit Schedule | 10<br>16 |
| 3.2 Testing Procedures | |
| STUDY PROCEDURES | |
| 4.1 Imaging Procedures | 1, |
| 4.2 Other Procedures | |
| MISCELLANEOUS CONSIDERATIONS | |
| 5.1 Treatment of DR and DME. | 18 |
| 5.2 Risks and Benefits. | |
| 5.3 Study Participant Withdrawal and Losses to Follow-up | |
| 5.4 Discontinuation of Study | |
| 5.5 Contact Information Provided to the DRCR.net Coordinating Center | |
| 5.6 Subject Reimbursement | |
| CTATICTICAL CONCIDED ATIONS | 20 |
| 6.1 Primary Outcome | |
| 6.2 Sample Size Estimation | |
| 6.3 Primary Analysis Plan | |
| 6.3.1 Principles for Analysis | |
| 6.3.2 Confounding | |
| 6.3.3 Per Protocol Analyses | |
| 6.3.4 Sensitivity Analyses | |
| 6.3.5 Subgroup Analyses | |
| 6.4 Secondary Outcomes and Safety Outcomes for Treatment Group Comparison | |
| DATA COLLECTION AND MONITORING | 2 <del>-</del> 7 |
| DATA COLLECTION AND MONITORING 7.1 Case Report Forms | 20<br>26 |
| 7.2 Study Records Retention | |
| 7.3 Quality Assurance and Monitoring | |
| 7.4 Protocol Deviations | |
| / I I I I I I I I I I I I I I I I I I I | / |

| ETHICS/PROTECTION OF HUMAN PARTICIPANTS | 28 |
|--------------------------------------------|----|
| 8.1 Ethical Standard | 28 |
| 8.2 Institutional Review Boards | 28 |
| 8.3 Informed Consent Process | 28 |
| 8.3.1 Consent Procedures and Documentation | 28 |
| 8.3.2 Participant and Data Confidentiality | 28 |
| REFERENCES | 30 |

# **ABBREVIATIONS**

| ACCORD | Action to Control Cardiovascular Risk in Diabetes |
|---|---|
| ACCORD-Eye | Action to Control Cardiovascular Risk in Diabetes Eye Trial |
| ALT | Alanine aminotransferase |
| anti-VEGF | Anti-Vascular Endothelial Growth Factor |
| AST | Aspartate aminotransferase |
| bid | Two times per day |
| CI | Confidence Interval |
| CK | Creatine kinase |
| CST | Central Subfield Thickness |
| DME | Diabetic Macular Edema |
| DR | Diabetic Retinopathy |
| DRCR.net | Diabetic Retinopathy Clinical Research Network |
| E-ETDRS | Electronic- Early Treatment Diabetic Retinopathy Study |
| ETDRS | Early Treatment Diabetic Retinopathy Study |
| FIELD | Fenofibrate Intervention and Event Lowering in Diabetes |
| HbA1c | Hemoglobin A1c |
| HR | Hazard Ratio |
| ICH | International Conference on Harmonization |
| IRB | Institutional Review Board |
| JCHR | Jaeb Center for Health Research |
| NF-kappa B | nuclear factor kappa-light-chain-enhancer of activated B cells |
| NPDR | Non-Proliferative Diabetic Retinopathy |
| OCT | Optical Coherence Tomography |
| PDR | Proliferative Diabetic Retinopathy |
| PPARα | Peroxisome Proliferator-Activated Receptor α |
| PROMINENT | Pemafibrate to Reduce Cardiovascular Outcomes by Reducing<br>Triglycerides in Patients with Diabetes |
| PRP | Panretinal Photocoagulation |
| QALY | Quality-Adjusted Life-Year |
| US | United States |
| UWF | Ultra-widefield |

#### 1.1 Diabetic Retinopathy Complications and Public Health Impact

The age-adjusted incidence of diabetes mellitus in the United States has reportedly doubled in recent history. Estimates suggest that by the year 2040, approximately 642 million individuals worldwide will be affected by this chronic disease. The increasing global epidemic of diabetes implies an increase in rates of associated vascular complications from diabetes. At present, almost 8 million people in the United States are estimated to have diabetic retinopathy (DR). Despite advances in the diagnosis and management of ocular disease in patients with diabetes, eye complications from diabetes mellitus continue to be a leading cause of vision loss and new onset blindness in working-age individuals throughout the United States. The increasing global epidemic of diabetes implies an increase in rates of associated vascular complications from diabetes. At present, almost 8 million people in the United States are estimated to have diabetes retinopathy (DR). Despite advances in the diagnosis and management of ocular disease in patients with diabetes, eye complications from diabetes mellitus continue to be a leading cause of vision loss and new onset blindness in working-age individuals throughout the United States.

# 1.2 Preventing DR Onset and Worsening

At this time, the primary method of slowing DR onset and worsening remains that of strict glycemic control and blood pressure control. Results from the Early Treatment Diabetic Retinopathy Study (ETDRS) revealed that better glycemic control inhibits DR worsening among all age groups, type 1 and type 2 diabetes, and all stages of retinopathy. The United Kingdom Prospective Diabetes Study (UKPDS) and the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Study demonstrated that improved blood glucose control can reduce the risk of developing DR in patients with type 2 diabetes, with the UKPDS additionally showing the benefit of improved blood pressure control.<sup>7,8</sup> The Diabetes Control and Complications Trial (DCCT) found that intensive therapy, aimed at keeping glycemic levels as close to normal range values as possible, reduced the risk of any DR developing by 76% (95% confidence interval (CI):62% to 85%) among patients with no DR at baseline and slowed the worsening of DR by 54% (95% CI: 39% to 66%) among patients with mild DR at baseline. The benefits of intensive treatment were sustained for approximately 4 years after the period of intensive glycemic control with a 75% (P<0.001) risk reduction in the worsening of DR. 10 This beneficial effect in fact persisted for even as long as 18 and 25 years later in this cohort of study participants with type 1 diabetes. <sup>11, 12</sup> This beneficial effect also persisted in type 2 diabetes. 13, 14

Despite improvements in systemic glycemic control, <sup>15</sup> there continues to be a substantial proportion of diabetic patients who develop DR and its associated sequelae. In 2005–2008, 28.5% (4.2 million) of Americans with diabetes aged 40 years or older had DR, and of this group, 655,000 individuals had advanced DR that could lead to severe vision loss. <sup>16</sup> Approximately 40-60% of the Wisconsin Epidemiologic Study Diabetic Retinopathy (WESDR) cohort, whose onset of diabetes occurred between 1922 and 1980, developed proliferative diabetic retinopathy (PDR) over time, with rates of visual impairment (vision of 20/40 or less in the better seeing eye) ranging from approximately 5% to 20%. <sup>15</sup>

#### 1.3 Limitations of Current Treatments for PDR and DME

Recent advances in therapy for advanced diabetic eye disease include the use of anti-vascular endothelial growth factor (anti-VEGF) agents to prevent vision loss from PDR and also to treat center-involved DME. Anti-VEGF therapy has been shown to be highly effective in treating active ocular neovascularization as well as in increasing visual gain and decreasing visual loss in eyes with center-involved DME. <sup>17-19</sup> However, anti-VEGF treatment does have drawbacks including the need for recurrent intravitreous injections for medication delivery that are performed as often as once a month. These injections have potential associated side effects including the development of endophthalmitis and incremental cost effectiveness ratios when using aflibercept or ranibizumab that are far beyond \$100,000 per Quality-Adjusted Life-Year (QALY) over a 10-year time horizon compared with bevacizumab. <sup>20</sup> In addition not all eyes treated with anti-VEGF have resolution of

DR or DME. 19, 21 Scatter laser photocoagulation or panretinal photocoagulation (PRP) is another treatment for PDR that is not invasive and does not need to be repeated as frequently as anti-VEGF injections, but laser treatment has other well-documented adverse effects, including exacerbation or development of macular edema with transient or permanent central vision loss, peripheral visual field defects, night vision loss, loss of contrast sensitivity, potential complications from misdirected or excessive burns, increased risk of vitrectomy compared with anti-VEGF treatment, and worsening of visual loss in nearly 5 percent of individuals despite appropriate treatment. <sup>19,22</sup> Thus. there is an ongoing need to identify novel therapies that are both effective for PDR and DME treatment and that also avoid the potential adverse events or costs associated with current ocular interventions. Furthermore, the identification of an oral therapeutic agent that may prevent worsening to PDR or DME might allow treatment of a wider segment of the diabetic population at risk for diabetic eve complications who do not have access to anti-VEGF or laser treatment or who are not suitable candidates for these treatments. This would be a major public health contribution if indeed this potentially effective oral agent could be implemented into clinical care.

# 1.4 Rationale for PPARa Therapy for DR Worsening

Two major clinical studies in patients with diabetes have demonstrated beneficial effects on ocular outcomes from treatment with oral fenofibrate, which acts via activation of peroxisome proliferator-activated receptor α (PPARα) and may decrease inflammation through inhibition of NF-kappa B activity. Fenofibrate is an oral medication of the fibrate class with a well-documented and favorable safety profile that is used for treatment of hyperlipidemia. Fenofibrate reduces low-density and very low-density lipoprotein and triglyceride levels while increasing high-density lipoprotein levels. In addition to its agonist effects on the PPARα pathway, fenofibrate affects human retinal endothelial cells through a PPARα-independent mechanism. A number of other pathways have also been explored with regards to its effects in diabetic retinopathy. For example, Dr. Lois Smith from Harvard has suggested that fenofibrate may inhibit cytochrome P450 epoxygenase 2C activity resulting in reduction in pathological ocular angiogenesis, using her oxygen induced retinopathy in a mouse model. Others have suggested a decrease in NF-kappa B activity may be the potential pathway for reduction of diabetic retinopathy progression. Other mechanisms have also been suggested.

The Fenofibrate Intervention and Event Lowering in Diabetes (FIELD) study randomized 9795 patients with type 2 diabetes to fenofibrate 200 mg/day versus placebo.<sup>30</sup> A subgroup of this cohort (N=1012) also agreed to undergo fundus photography at baseline, 2 year, 5 year, and end of study in order to document DR severity worsening. The percentage of patients requiring first laser treatment for either DR or DME was significantly lower in the fenofibrate group than in the placebo group (3.4% vs 4.9%; HR for first laser treatment: 0.69, 95% CI 0.56-0.84, P = 0.0002). 850 participants (84%; 421 allocated to placebo, 429 allocated to fenofibrate) in the photography substudy were followed to the end of the study. Although a difference between the groups overall for the primary endpoint of 2-step DR worsening in the substudy was not identified, in the subgroup of participants with pre-existing DR (N=193), fenofibrate treatment was associated with a reduction in 2-step DR worsening as compared with placebo (3.1% versus 14.6%, P = 0.004).

The Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial enrolled 10,251 participants with type 2 diabetes and randomized them to intensive glycemic control (goal HbA1c < 6.0%) or standard therapy. The 5,518 participants with dyslipidemia were further randomized in a 2x2 factorial design to receive simvastatin in combination with either fenofibrate (at 160 or 54 mg/day depending on renal function) or placebo. The ACCORD Eye study enrolled 3,537 individuals from this group of which 82.3% (N = 2,856) achieved both a baseline and year 4 follow-up visit and among which 1,593 were included in the fenofibrate portion of the trial. Among all of

the participants in the ACCORD Eye trial, 1,370 (48%) had no diabetic retinopathy in either eye, 892 (31%) had mild diabetic retinopathy, 553 (19%) had mild to moderately severe NPDR, and 39 (1%) had severe NPDR or PDR (note: 2 participants were not classified).

At 4 years, DR worsening was significantly less likely with intensive glycemic control as compared with standard therapy (7.3% vs. 10.4%; adjusted OR, 0.67, 95% CI, 0.51-0.87, P = 0.003). DR worsening also was significantly less frequent in the fenofibrate as compared with the placebotreated group (6.5% versus 10.2%, adjusted OR, 0.60, 95% CI, 0.42-0.87, P = 0.006). The benefit of fenofibrate therapy was seen primarily in study participants with DR at baseline (see table below). In patients with microaneurysms in only 1 or both eyes or with mild nonproliferative diabetic retinopathy (NPDR) in only 1 eye, the odds ratio for >3 step progression was 0.27 (95% CI: 0.12-0.63, p = 0.0009). No significant relationship was seen between fenofibrate use and DR worsening in eyes with no DR. Among participants with mild NPDR to moderately severe NPDR (N = 279) the rates of progression were 9% to 17%. Fenofibrate treatment did not appear to affect the rate of at least moderate vision loss (fenofibrate group: 23.7%, vs. placebo group: 24.5%, P = 0.57), nor did it affect changes in macular edema status between baseline and year 4.

| Tools : | True Non | e frame of Track | esta Dante da sel | e known | memulan Sama | Land in Schengers |
|---|---|---|---|---|---|---|
| 1.1.740 3. | 11 74 FT + 3 6 2 | P. I. CARNID CONTRACTOR | ALTO INVESTIGATION | The Property of the Control of the C | DESCRIPTION OF STREET | PROPERTY AND PROPERTY |

| | Hyenna Tesi | | | light Teil | | | Physil Pressure Trial | | |
|---|---|---|---|---|---|---|---|---|---|
| Chitoroph | bank | Services | 05 (15% 10) | * English | Cash | 241 (49,542, 7 | head.c | hoded | 08,994030,4 |
| Origina sout of a coversouse<br>(21 cm - PC or sound as) | | 2304 ( 40/46) | 057(05 DM)<br>7 = 00775 | DOM: (52/88) | (000,000%) | 1080 (0.42 Gest)<br>P = 0.0006 | | 1766 (566); | ta: 0.84 0.9<br>P = 2.39 |
| Kesterland sidepagement<br>(2) explor PC) | 2008 (45,0455) | \$357 (14V 457) | 2014 (0.42-0.14)<br>P = 0.440 | 19361 (45406) | 1936-(52/56) | P = 0.0019 | DARK (MAN) | 019 4 (57,90%) | P = 0.33 |
| Inchasig Lincoln | 2003 (35063) | 120 HAX 571 | 071-051-30<br>7 027 | 0.063 (35+01) | 0030132070 | F 0.72 | 2,002 (21/27) | 1.040 (52/282) | 1 0000 V -1 40 |
| Backing resp. 2 (A) Ma<br>on the MICO Section 13<br>on Na only in tilture | 2027 (12935) | . 354 (98)(59) | 09: (VL) 138/<br>V 079R | 0.030 (\$100) | | 0.27 (0.12 × 60)<br>P = 7000W | 2005 (2017) | COLUMN | 1.12 (0.00 - 5.40<br>P = 0.71 |
| basel ne west to A.<br>millionskene NPOR | 5080 (58910) | 2313 (20) (21) | 7 = 0.75 | 1000 10460 | 30155 (14/404) | Ref (0.0+1 15)<br>P = 0.79 | 2.Mr. (5.64) | Called (Ma) | 190 BGS - 1.50<br>P = 2.33 |
| finel matery 7–9<br>replaced made and<br>serve NIDE | 2.04 (1753) | 230 (2004) | 5 = 5.49<br>0.34 (0.32+1.85) | AD4-09-71 | 0.00000 | P = 0.21 | 1201 ( M) | 2.222 (5900) | 2.37 (246—7.24<br>P = 3.30 |
| Noting and 10. In own.<br>NOTE: 733 | 1999 (12/15) | 2583 ( 4/240 | 10 | (1/0%) (4-5) | 28 640 | | 0.006 (1.00%) | 28.186 | |
| AULAND - Action to Compel C<br>patient for damping and property<br>face left in the form prompty<br>M. Hell I - a compel to make | Separate. | | facete iutoczeny | , Ha • ri zvero | arsevi NULL | nonproliferative a | libete vernopat | ng Kili pheno | vytaka 1500 |

\*Table taken from Chew EY, Davis MD, Danis RP, et al. The effects of medical management on the progression of diabetic retinopathy in persons with type 2 diabetes: the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Eye Study. *Ophthalmology*. 2014;121(12):2443-51.

In the 8 year follow-up study of ACCORD, 4 years following the cessation of the fenofibrate, the rates of diabetic retinopathy progression was 11.8% (47 of 399) in the fenofibrate group and 10.2% (37 of 363) in the placebo group with an adjusted odds ratio (OR) of 1.13 (95% CI: 0.71-1.79; P =0.60), suggesting the benefit does not persist once the drug is stopped. Using the Cox proportional hazards model resulted in an adjusted HR of 0.76 (95% CI 0.57-1.03, P = 0.08). When adjusted for the competing risk of death, the adjusted HR was 0.83 (95% CI 0.69-1.00, P = 0.04).  $^{14}$ 

# 1.5 Pemafibrate and the Ongoing PROMINENT trial

Pemafibrate is a highly selective and potent modulator of PPARα. Pemafibrate, a selective peroxisome proliferator alpha receptor modulator (SPPARM-α), is approximately 2,500 times more potent than fenofibric acid, in terms of the concentration, producing 50% effectiveness (i.e., effective concentration in 50% of participants [EC<sub>50</sub>]) of the PPARα-activating effect. The Pemafibrate to Reduce Cardiovascular Outcomes by Reducing Triglycerides in Patients with Diabetes (PROMINENT) study is a phase 3 multinational, multicenter, randomized, placebocontrolled masked trial to assess whether treatment with pemafibrate will delay the time to occurrence of the composite cardiovascular outcome of nonfatal myocardial infarction, nonfatal

ischemic stroke, unstable angina requiring unplanned revascularization and/or cardiovascular death. The participants are adults with type 2 diabetes who have elevated triglycerides and low high-density lipoprotein cholesterol, and are at high risk for cardiovascular events, in the context of adequate background of lipid-lowering therapy (including stable dose moderate or high intensity statin). Two-thirds of the enrolled study population will have prior evidence of systemic atherosclerosis (secondary prevention cohort) while one-third will not (high risk primary prevention cohort, age  $\geq 50$  years [male] or  $\geq 55$  years [female]). There are expected to be approximately 2,500 participants enrolled in the U.S. and Canada. The trial is an event-driven trial, anticipated to involve approximately 10,000 participants to achieve 1,092 cardiovascular events over approximately 5 years.

This protocol is an ancillary study to the main PROMINENT trial in which the DRCR.net and PROMINENT Study Group will collaborate to evaluate the effect of pemafibrate treatment versus placebo on long-term rates of DR worsening in patients with type 2 diabetes at risk for cardiovascular events. Based on data from eyes with baseline retinopathy in the ACCORD Eye study (see table below), it is anticipated that approximately 50% of PROMINENT study participants will have diabetic retinopathy in at least one eye and be eligible for this PROMINENT-Eye Study.

Table 2. Bue the Challe Chapteris in all ACCARD Ep. Survey.

For existents.

| Characteristics | No. Penkipun<br>1%) |
|---|---|
| Boseline severity of discretic setting only | SO CHARKS |
| None Corel 10, mer 11 | 1370 (48.0) |
| Micromanyous only Heads 20 (22), steps 2 (3) | 308 (21.0) |
| khal NP.X. (heads 25 ≤35, steps 1-5) | 559 (19.9) |
| M. Jeute N. UK (leves 42545), v.e., 6-77 | 125 (6.2) |
| Mindewrels were KTDS (less s 47.047)<br>sees 8-49 | 101 (3.5) |
| Service N. USC (PAR (feve. 55-57) in 4 mass., steps. 10, 17) | 39 (2.4) |
| Magalar cilona (2005e eye) | |
| None (LLD0.5 LME revening CA) | 25/9 (95.1) |
| Mtd (tB-(C) | 159 (5.3) |
| Medicani (2 - 370) | 44 (7.5) |
| Several (mmSC) | 25 (3.5) |
| Load enables also total [4] person. | |
| Name (C.DA.) | 2500 (90.7) |
| Vey mid to 0 and < 0.0 hi Dot | 117.76.16 |
| Mid (20.016 and <0.127 DA) | 128 3651 |
| Moderate (≥0.125 DAS | 23 (3.7) |
| Social thickening to along person. | |
| Name (C.DA) | 3421 (91.9) |
| Very mild (a Cond a 0.49 DA) | 55 (3.3) |
| Mid (3 C / 0 and < 1,50 DA) | 75-72,64 |
| Maderate (>1.99 and <0.25 EW) | 49.71.70 |
| Serce (262) UA: | 12 (0.4) |
| ACCRC = Action to Control Codics and Ir Rich<br>disc uses EIDSS - Early Transacte Dislocate<br>SAUR = Locapo literative deleta sette policy IV | artisignity. South |

Table taken from Chew EY, Davis MD, Danis RP, et al. The effects of medical management on the progression of diabetic retinopathy in persons with type 2 diabetes: the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Eye Study. *Ophthalmology*. 2014;121(12):2443-51.

#### 1.6 Summary of Protocol Rationale

Despite improved glycemic and systemic control for many patients with diabetes, over the past several decades, DR develops and progresses in a large proportion of patients, and visual loss from diabetic eye complications continues to be a leading cause of blindness in the US and other developed countries worldwide. Thus, even a modest ability to prevent DR onset or to slow DR worsening might substantially reduce the number of patients at risk for diabetes-related vision loss

worldwide. Widespread use of an oral agent effective at reducing worsening of DR might also 167 168 decrease the numbers of patients who undergo treatment for DR and DME and who are 169 consequently at risk for side effects that adversely affect visual function. Two major studies of 170 fenofibrate, FIELD and ACCORD-eye, have demonstrated clinically important reduction in 171 progression of retinopathy in patients with diabetes assigned to fibrate compared with placebo. 172 However, despite the positive clinical trial results, fenofibrate has not gained wide acceptance as a 173 preventive agent by either ophthalmologists or primary diabetes care providers. Thus, it is 174 important to provide further evidence demonstrating whether or not selectively increasing PPARa 175 activity reduces progression of retinopathy in patients with diabetes and non-proliferative diabetic retinopathy at baseline. Pemafibrate is a more potent and selective PPARα modulator than 176 177 fenofibrate. Its efficacy is currently being evaluated in the PROMINENT study for prevention of 178 cardiovascular events in patients with type 2 diabetes. Given the large study cohort with a 179 substantial proportion likely to have DR and the multi-year duration of the PROMINENT trial, this 180 study represents a unique opportunity to assess effects of chronic PPARa activation through 181 pemafibrate therapy on DR outcomes.

182 183

# 1.7 Study Objective

184 185

186

187

188

# **Primary Objective:**

1. To assess whether treatment with pemafibrate (0.2 mg orally BID) compared with placebo reduces the hazard rate of diabetic retinopathy worsening in adults with type 2 diabetes and

diabetic retinopathy without neovascularization in at least one eye who are participating in the parent PROMINENT trial.

189 190 191

### **Secondary Objectives:**

193 194

192

1. To assess whether treatment with pemafibrate (0.2 mg orally BID) compared with placebo reduces rates of diabetic macular edema development or visual acuity worsening.

195 196

2. To assess whether treatment with pemafibrate compared with placebo affects safety or tolerability in the cohort of participants with diabetic retinopathy in at least one eye.

197 198

199

### 1.8 Study Design and Synopsis of Protocol

# A. Study Design

• Longitudinal ancillary study to the PROMINENT trial.

200 201 202

# B. Major Eligibility Criteria (see section 2.2 for additional eligibility criteria)

203

• Already randomized at US or Canadian sites in the PROMINENT study

204 205 a. Enrollment visit into the ancillary study must be conducted within 3 months of randomization into the PROMINENT trial.

206 207 • Ability to cooperate with dilated ophthalmic examination and imaging procedures • At least one eye meets the following study eye inclusion criteria:

208 209 a. ETDRS Diabetic Retinopathy Severity level between 20 and 53 (minimal to severe NPDR), inclusive, according to the investigator and confirmed by central Reading Center grading.

210 211

Major study eye exclusion criteria are:

212 213 a. Neovascularization on clinical exam or fundus photographs b. Current central-involved DME based on optical coherence tomography (OCT) central subfield thickness (CST)

214 215

- i. Zeiss Cirrus:  $CST \ge 290 \mu m$  in women or  $\ge 305 \mu m$  in men
- ii. Heidelberg Spectralis: CST  $\geq 305 \mu m$  in women or  $\geq 320 \mu m$  in men

- c. Major non-diabetic intraocular pathology that in the opinion of the investigator would substantially and adversely affect visual acuity or lead to ocular neovascularization during the course of the study
- d. Anticipated need for intravitreous anti-VEGF, intravitreous corticosteroid, or PRP in the next 6 months following randomization
- e. History of intravitreous anti-VEGF or corticosteroid treatment within the prior year for any indication.
- f. Any history of PRP or vitrectomy

Participants may have 1 or 2 study eyes based on how many eyes meet eligibility criteria.

### C. Estimated Sample Size

At least 600 individuals are expected to be eligible and to enroll in the study at US and Canadian DRCR.net clinical sites that have geographic proximity to the parent PROMINENT clinical site. Recruitment will continue until the PROMINENT trial has completed enrollment, with up to a maximum of 900 enrolling in PROMINENT-Eye.

# **D.** Protocol Summary

Participants in the parent PROMINENT study will be referred to partnering DRCR.net sites for comprehensive ophthalmologic examination including visual acuity, fundus photography and spectral domain optical coherence tomography (OCT) to be performed within 3 months of the PROMINENT randomization visit. Participants who meet eligibility criteria at this visit will be eligible for two or three additional study ophthalmic visits through 4 years (see Table in Section E below). Participants who do not meet ocular eligibility will be discontinued from the ancillary PROMINENT-Eye Study, but not from the parent study. If intravitreous anti-VEGF or corticosteroid treatment, PRP, or vitrectomy will be administered to a study eye for any indication for the first time since entering the study, when possible, all study procedures should be performed prior to implementing treatment to establish retinopathy severity before therapy is initiated. Participants who receive treatment will continue follow-up through 4 years.

# E. Schedule of Study Visit and Examination Procedures

| Visit and Visit Window | Screening/<br>Baseline <sup>a</sup> | 2 year <sup>b</sup><br>± 2 months | 4 year <sup>b</sup><br>± 2 months <sup>c</sup> | Prior to<br>DME/PDR<br>Treatment<br>Initiation <sup>d</sup> |
|---|---|---|---|---|
| Best corrected visual acuity | X | X | X | X |
| Eye Exam <sup>e, f</sup> | X | X | X | X |
| DRCR.net Fundus<br>Photography <sup>e,g</sup> | X | X | X | X |
| Spectral Domain OCT <sup>e</sup> | X | X | X | X |
| Collection of Adverse<br>Events occurring during<br>the visit | X | X | X | X |

- a. To be performed within 3 months of the PROMINENT randomization visit
- b. Time from randomization into the PROMINENT trial.

- c. If the PROMINENT trial ends before a participant reaches the 4 year visit, one final visit within 3 months of
   the PROMINENT trial ending will be completed.
- d. All study procedures should be performed prior to the initiation of treatment for DME or DR in a study eye.
- e. After pupil dilation
  - f. Participants may opt out of eye exam particularly if they have recently had an eye exam
  - g. The widest camera type available will be used for color fundus photography.

# F. Outcomes

#### Primary outcome:

The primary outcome is diabetic retinopathy worsening or DME development (composite outcome), based on both eyes for bilateral participants and based on the study eye only for unilateral participants. Study eye is defined based on the criteria in section 2.2.2 as the eye(s) having ETDRS Diabetic Retinopathy Severity level between 20 and 53 (minimal to severe NPDR), inclusive, according to the investigator and confirmed by central Reading Center, without definite central subfield involved diabetic macular edema.

Diabetic retinopathy worsening or DME development is defined as any of the following:

- For participants with 2 study eyes: 3-step worsening on the ETDRS Retinopathy Severity Scale for Persons (Table 1 in Section 6) at a protocol visit. This scale takes into account the retinopathy level of both study eyes.
- For participants with one study eye: 2-step worsening on the ETDRS Retinopathy Severity Scale for Individual Eyes (Table 2 in Section 6) in the study eye at a protocol visit. This scale only takes into account the retinopathy level of the study eye.
- Procedure undertaken for the treatment of PDR at any time (even in the absence of photographic documentation) including PRP, intravitreous anti-VEGF, or vitrectomy in at least one study eye.
- Treatment initiated for DME at any time (even in the absence of OCT documentation) including anti-VEGF, corticosteroids, focal/grid laser, or vitrectomy in at least one study eye.
- Development of central-involved DME on OCT with vision loss at the 2-year or 4-year visit. Defined as OCT central subfield thickness above the machine and gender-specific thresholds (see Section 2.2.2 for details) with at least a 10% increase in thickness from baseline and visual acuity 20/32 or worse (letter score ≤ 78) in at least one study eye.

Secondary outcomes include a treatment comparison of the following:

<u>Participant-Level Secondary Outcomes (relates to either eye for bilateral participants and to the study eye for unilateral participants):</u>

- Hazard rate of 3-step person-level (for bilateral participants, see Table 1 in Section 6) or 2-step eye-level (for unilateral participants, see Table 2 in Section 6) diabetic retinopathy worsening on the ETDRS Retinopathy Severity Scale or receiving treatment for PDR in at least one study eye at any time (irrespective of DME status or treatment)
- Hazard rate of developing central-involved DME on OCT with vision loss (as defined above) or receiving treatment for DME in at least one study eye at any time (irrespective of diabetic retinopathy severity level or treatment)
- Person-level diabetic retinopathy severity at 2 years and 4 years
- Percentage of participants with at least a 2-line loss in visual acuity from baseline in at least one study eye at 2 years and 4 years

**Eye-Level Secondary Outcomes** (evaluated only for study eyes):

302303

304

305306

307

308

309

310

311312

313

314315

316

- Hazard rate of a composite PDR/DME outcome. Defined as the time to 2-step diabetic retinopathy worsening on the ETDRS Retinopathy Severity Scale for Individual Eyes (see Table 2 in Section 6) at 2 years or 4 years, development of central-involved DME on OCT with vision loss (as defined above) at 2 years or 4 years, or treatment for DME or PDR at any time
- Hazard rate of 2-step diabetic retinopathy worsening or receiving treatment for PDR at any time (irrespective of DME status or treatment)
- Hazard rate of developing central-involved DME on OCT with vision loss at 2 years or 4 years or receiving treatment for DME at any time (irrespective of diabetic retinopathy level or treatment)
- Eye-level diabetic retinopathy severity at 2 years and 4 years
- Change in OCT central subfield thickness from baseline at 2 years and 4 years
- Change in visual acuity letter score from baseline at 2 years and 4 years
- Percentage of eyes with at least 2-line loss in visual acuity from baseline at 2 years and 4 years

317318319

320

321

#### Safety Outcomes:

- Adverse events collected as part of this ancillary study including vitreous hemorrhage and retinal detachment
- Changes from randomization in ALT, AST, CK, and creatinine

322323324

325

326327

#### 1.9 General Considerations

The study is being conducted in compliance with the policies described in the DRCR.net Policies document, with the ethical principles that have their origin in the Declaration of Helsinki, with the protocol described herein, and in accordance with ICH E6 Good Clinical Practice. All study investigators will attest to complying with these requirements.

328 329 330

The DRCR.net Procedures Manuals provide details of the imaging procedures.

331332

Retinal images and OCT data will be primary source data, and additional data collected will be directly entered in electronic case report forms, which will be considered the source data.

333334

There is no restriction on the number of participants to be enrolled by a site.

335336

Assessment of adverse events occurring during the Prominent-Eye clinical visit will be obtained through adverse event reporting at the end of each study visit.

339

A risk-based monitoring approach will be followed, consistent with the FDA "Guidance for Industry Oversight of Clinical Investigations — A Risk-Based Approach to Monitoring" (August 2013).

343

344 The risk level for this ancillary research is considered to be no more than minimal risk.

#### STUDY PARTICIPANT ELIGIBILITY AND ENROLLMENT

345 346 347

348

349

350

351

352

353 354

355

356

357

### 2.1 Identifying Eligible Participants and Obtaining Informed Consent

At least 600 participants are expected to be enrolled in this study. Recruitment will continue until the PROMINENT trial has completed enrollment, with up to a maximum of 900 participants enrolling in PROMINENT-Eye. Participants in the PROMINENT trial will be referred to participating DRCR.net sites based on geographic proximity within the U.S. and Canada. The ancillary study brochure providing an overview of the study will be initially discussed with the patient by the PROMINENT investigator and/or coordinator. Interested participants will be provided contact information and encouraged to contact their local PROMINENT-Eye clinical site and (if permitted by the IRB) will consent to having their contact information provided to the local PROMINENT-Eve clinical site and the DRCR.net Coordinating Center. The DRCR.net PROMENENT-Eye clinical site may also contact the participant to facilitate scheduling with participant consent.

358 359 360

361

362

363

364

At the DRCR.net clinical site, the PROMINENT-Eye study protocol will be discussed with the patient by a DRCR.net study investigator and clinic coordinator. Prior to completing any procedures or collecting any data for this study, informed consent will be obtained. Potential eligibility will be assessed at the screening visit. Patients who are eligible based on the screening visit and Reading Center confirmation of DR severity level will return for additional study imaging visits as outlined below.

365 366 367

368 369

370

371

#### 2.2 Subject Eligibility and Exclusion Criteria

# 2.2.1 Eligibility Criteria

- Already randomized at US or Canadian sites in the PROMINENT study
  - a. Enrollment visit into the ancillary study must be conducted within 3 months of randomization into the PROMINENT trial.
- Ability to cooperate with dilated ophthalmic examination and imaging procedures

372 373 374

#### 2.2.2 Study Eye Criteria:

The study participant must have at least one eye meeting all of the inclusion criteria listed below.

375 376 377

The eligibility criteria for a study eye are as follows (both eyes will be considered study eyes if both meet the eligibility criteria at the time of enrollment):

378 379 380

• At least one eye meets the following study eye inclusion criteria:

381 382 a. ETDRS Diabetic Retinopathy Severity level between 20 and 53 (minimal to severe NPDR), inclusive, on color fundus photographs confirmed by central Reading Center grading.

383 384

• Study eye exclusion criteria are:

a. Neovascularization present.

385 386

b. Current central-involved DME based on optical coherence tomography (OCT) central subfield thickness (CST)

387 388

i. Zeiss Cirrus: CST  $\geq$  290µm in women or  $\geq$  305µm in men ii. Heidelberg Spectralis: CST  $\geq 305 \mu m$  in women or  $\geq 320 \mu m$  in men

389

c. Known major non-diabetic intraocular pathology that in the opinion of the investigator would substantially and adversely affect visual acuity or lead to ocular neovascularization during the course of the study

390 391

- d. Anticipated need for intravitreous anti-VEGF, intravitreous corticosteroid, or PRP in the next 6 months following randomization
  - e. History of intravitreous anti-VEGF or corticosteroid treatment within the prior year for any indication.
  - f. History of intraocular surgery within prior 4 months or anticipated within the next 6 months following randomization
  - g. Any history of PRP or vitrectomy
  - h. History of YAG capsulotomy performed within 2 months prior to screening
  - i. Aphakia
  - j. Known substantial media opacities that would preclude successful imaging

Participants may have 1 or 2 study eyes based on how many eyes meet eligibility criteria.

404 405 406

407

408

395396

397398

399

400 401

402

403

## 2.3 Screening Evaluation and Baseline Testing

#### 2.3.1 Ocular Historical Information

An ocular history will be elicited from the potential study participant including prior ocular diseases, surgeries, and treatment.

409 410 411

412

413

414

415

416

417

418

# **2.3.2 Baseline Testing Procedures**

The following procedures will be performed to assess eligibility and/or to serve as baseline measures for the study:

- The testing procedures are detailed in the DRCR.net Procedures Manuals. Visual acuity testing, ocular exam, fundus photography, and OCT will be performed by DRCR.net certified personnel.
- The fundus photographs will be sent to a Reading Center for grading.
- OCT images meeting DRCR.net criteria for manual grading will be sent to a Reading Center.

419 420

- 1. E-ETDRS visual acuity testing at 3 meters using the Electronic Visual Acuity Tester (including protocol refraction) in each eye
- 423 2. Ocular examination on each eye including dilated ophthalmoscopy
  - Participant can opt out of ocular exam (dilation will be required regardless)
- 425 3. Spectral Domain OCT using Zeiss Cirrus or Heidelberg Spectralis OCT machine on both eyes
- 426 4. DRCR.net protocol fundus photography in both eyes
- The widest field camera type available will be used for color fundus photography.

#### FOLLOW-UP VISITS

# 428 429

430

#### 3.1 Visit Schedule

Each participant will have protocol specific follow-up visits scheduled at 2 years ( $\pm$  2 months) and at 4 years ( $\pm$  2 months) from the randomization date in the PROMINENT trial. If the

PROMINENT study ends prior to a participant's 4-year visit, the participant will have one closeout visit within 3 months of the last PROMINENT visit.

434 435 436

437

438

439

440

441

442

443

444

445

433

Additional retina evaluation visits may occur as required for usual care of the study participant either by the DRCR.net clinical site or by the participant's non-DRCR.net ophthalmologist. If the participant will be examined by a non-DRCR.net ophthalmologist, the participant will be asked to sign a medical records release so any treatment that is documented can be obtained by the DRCR.net site. In addition, participants for whom ocular treatment for DR or DME is planned for the first time during the trial (e.g. anti-VEGF or corticosteroid intravitreous injection, PRP, focal/grid laser, or vitrectomy) will be asked to return to the DRCR.net clinical site to complete the study procedures before the treatment is administered, provided treatment is not urgently needed as determined by the treating physician. If pre-treatment images are not able to be obtained, study images should try to be obtained within 1 month after treatment initiation. Participants who receive

446 447 448

Communication between the PROMINENT clinical site and the PROMINENT-Eye clinical site may occur to facilitate compliance with the follow-up schedule if needed.

449450451

### 3.2 Testing Procedures

The following procedures will be performed at each protocol visit unless otherwise specified. A grid in section 1.3 summarizes the testing performed at each visit.

454

459

- 455 1. Visual Acuity:
- A protocol refraction followed by E-ETDRS visual acuity testing in both eyes (best corrected).
- 458 2. Ocular examination on each eye including dilated ophthalmoscopy
  - Participant can opt out of ocular exam (dilation will be required regardless)
- 460 3. OCT using Zeiss Cirrus or Heidelberg Spectralis OCT machine on both eyes
- 4. DRCR.net protocol fundus photography in both eyes

treatment will continue follow-up through 4 years.

• The widest field camera type available will be used for color fundus photography.

463

462

All of the testing procedures do not need to be performed on the same day, provided that they are completed within the time window of a visit and prior to initiating any treatment.

#### STUDY PROCEDURES

#### 4.1 Imaging Procedures

The DRCR.net protocol images will be obtained by a fundus photographer specifically certified by the DRCR.net for these imaging procedures. The images will be first sent to the DRCR.net Coordinating Center (uploaded through the website as available) and then to a Reading Center for further evaluation. During image grading, a map of the ETDRS 7 standard fields will be placed as an overlay on each ultra-widefield (UWF) image with peripheral areas outside the ETDRS fields darkened so that extent and severity of DR lesions can be graded separately for the areas within and outside the ETDRS fields.

OCT will be performed by DRCR.net certified personnel. Only spectral domain machines are permitted. For a given study participant, the same machine type should be used for the duration of the study, unless circumstances do not permit (e.g., replacement of damaged machine). If a switch is necessary, the same machine type should be used for the remainder of the study. The images will be sent to the DRCR.net Coordinating Center (uploaded through the website as available) and may be sent to a Reading Center for further evaluation.

Each digital image must be evaluated to be of adequate quality for submission, according to the study procedures. If photograph quality is judged substandard by the operator, then the imaging should be repeated until a good quality image is obtained.

#### **4.2 Other Procedures**

Ocular historical information will be collected, including prior treatment for diabetic retinopathy, prior nondiabetic ocular diseases, surgeries, and treatment.

#### 4.3 Safety Assessments

Assessment of subject safety at the study visit will be obtained through adverse event reporting at the end of each study visit. Any adverse events that occurred during the participant's visit will be documented and communicated to the PROMINENT clinical site, and these adverse events will be entered into the PROMINENT study database.

#### MISCELLANEOUS CONSIDERATIONS

#### 5.1 Treatment of DR and DME

Treatment of diabetic retinopathy and/or DME including initiation of PRP or anti-VEGF treatment is at the discretion of the treating physician. However, the first time PRP, intravitreous anti-VEGF or corticosteroid treatment, focal/grid laser, or vitrectomy is planned, the study procedures should be performed prior to treatment initiation, provided treatment is not urgently needed as determined by the treating physician.

#### 5.2 Risks and Benefits

The procedures in this study are part of daily ophthalmologic practice in the United States and pose few known risks. Dilating eye drops will be used as part of the exam. There is a small risk of inducing a narrow-angle glaucoma attack from the pupil dilation. However, all participants will have had prior pupil dilation usually on multiple occasions and therefore the risk is extremely small. Fundus photographs have bright lights associated with the camera flashes, which can be uncomfortable for study participants, but these carry no known risk to the eye or vision.

There may be few direct benefits from participating in this ancillary study other than the awareness of being involved in a large endeavor to answer relevant and timely questions regarding the possible benefit of pemafibrate on diabetic retinopathy progression.

In addition, if proliferative diabetic retinopathy is identified on color fundus photos, the participant's non-DRCR.net ophthalmologist (if applicable) and the PROMINENT investigator will be notified of this diagnosis so that treatment can be initiated if necessary.

#### 5.3 Study Participant Withdrawal and Losses to Follow-up

A study participant has the right to withdraw from the study at any time. If a study participant is considering withdrawal from the study, the principal investigator should personally speak to the individual about the reasons, and every effort should be made to accommodate him or her.

The goal for the study is to have as few losses to follow-up as possible. The Coordinating Center will assist in the tracking of study participants who cannot be contacted by the site. The Coordinating Center will be responsible for classifying a study participant as lost to follow-up.

Study participants who withdraw will be asked to have a final closeout visit at which the testing described for the protocol visits will be performed.

#### **5.4 Discontinuation of Study**

The study may be discontinued by the Executive Committee of the parent PROMINENT study or the Executive Committee of the PROMINENT-Eye study prior to the preplanned completion of follow-up for all ancillary study participants.

#### 5.5 Contact Information Provided to the DRCR.net Coordinating Center

The Coordinating Center will be provided with contact information for each study participant.
Permission to obtain such information will be included in the Informed Consent Form from the
PROMINENT study and from the PROMINENT-Eye study. The contact information will be
maintained in a secure database and will be maintained separately from the study data.

Contact from the Coordinating Center may be made for each study participant in the first month after enrollment, and approximately every six months thereafter. Additional contacts from the

- Coordinating Center will be made if necessary to facilitate the scheduling of the study participant for follow-up visits. A participant-oriented newsletter may be sent once a year. A study logo item may be sent once a year.
- 551 Study participants may be provided with a summary of the study results in a newsletter format after 552 completion of the study by all participants.
- 554 5.6 Subject Reimbursement
- The Coordinating Center will provide each study participant with a \$50 merchandise or money card per completed protocol visit. Additional travel expenses may be paid in cases for participants with
- higher expenses.

#### STATISTICAL CONSIDERATIONS

558 559 560

The approach to sample size and statistical analysis is summarized below. A detailed statistical analysis plan will be written and finalized prior to the completion of the study.

561 562 563

564

565 566

567

# **6.1 Primary Outcome**

The primary outcome is diabetic retinopathy worsening or DME development (composite outcome), based on both eyes for bilateral participants and based on the study eye only for unilateral participants. From a statistical perspective, the primary outcome is a person-level outcome as data from both eyes of bilateral participants is combined into a single outcome measurement. The primary outcome is defined as any of the following:

568 569 570

571

572

573

574

575 576

577

578

579 580

581

582

- For participants with 2 study eyes: 3-step worsening on the ETDRS Retinopathy Severity Scale for Persons (**Table 1**) at a protocol visit. This scale takes into account the retinopathy level of both study eyes.
- For participants with one study eye: 2-step worsening on the ETDRS Retinopathy Severity Scale for Individual Eyes (**Table 2**) in the study eye at a protocol visit. This scale only takes into account the retinopathy level of the study eye.
- Procedure undertaken for the treatment of PDR at any time (even in the absence of photographic documentation) including PRP, intravitreous anti-VEGF, or vitrectomy in at least one study eye.
- Treatment initiated for DME at any time (even in the absence of OCT documentation) including anti-VEGF, corticosteroids, focal/grid laser, or vitrectomy in at least one study eye.
- Development of central-involved DME on OCT with vision loss at the 2-year or 4-year visit. Defined as OCT central subfield thickness above the machine and gender-specific thresholds (see Section 2.2.2 for details) with at least a 10% increase in thickness from baseline and visual acuity 20/32 or worse (letter score  $\leq$  78) in at least one study eye.

583 584 585

586

Table 1: Summary of ETDRS Final Retinopathy Severity Scale for Persons

**Description** 

| 10/10 |
|---------|
| 20/< 20 |
| 20/20 |
| 35/< 35 |
| 35/35 |
| 43/< 43 |
| 43/43 |
| 47/< 47 |
| 47/47 |
| 501.50 |

Level in each eve

No DR

| 10/10 | NO DR | 1 |
|-------------------|---------------------------------------|----|
| 20/< 20 | Microaneurysms only, one eye | 2 |
| 20/20 | Microaneurysms only, both eyes | 3 |
| 35/< 35 | Mild NPDR, one eye | 4 |
| 35/35 | Mild NPDR, both eyes | 5 |
| 43/< 43 | Moderate NPDR, one eye | 6 |
| 43/43 | Moderate NPDR, both eyes | 7 |
| 47/< 47 | Moderately severe NPDR, one eye | 8 |
| 47/47 | Moderately severe NPDR, both eyes | 9 |
| 53/< 53 | Severe or very severe NPDR, one eye | 10 |
| 53/53 | Severe or very severe NPDR, both eyes | 11 |
| 60 or 61/< 60 | Mild PDR and/or PRP, one eye | 12 |
| 60 or 61/60 or 61 | Mild PDR and/or PRP, both eyes | 13 |
| 65/< 65 | Moderate PDR, one eye | 14 |
| 65/65 | Moderate PDR, both eyes | 15 |
| 71+/< 71 | High-risk PDR, one eye | 16 |
| 71+/71+ | High-risk PDR, both eyes | 17 |

587

Scale step

Table 2: Summary of ETDRS Final Retinopathy Severity Scale for Individual Eyes

| Level in the eye | Severity | Scale Step |
|---|---|---|
| 10 | DR absent | 1 |
| 20 | Microaneurysms only | 2 |
| 35 | Mild NPDR (hard exudates, soft exudates, and/or mild | 3 |
| | hemorrhage) | |
| 43 | Moderate NPDR (mild intraretinal microvascular abnormalities | 4 |
| | or moderate hemorrhage) | |
| 47 | Moderately severe NPDR (mild venous beading, moderate | 5 |
| | intraretinal microvascular abnormalities or severe hemorrhage) | |
| 53 | Severe or very severe NPDR (moderate/severe venous beading, | 6 |
| | severe intraretinal microvascular abnormalities and/or very | |
| | severe hemorrhage) | |
| 60, 61 | Scars of photocoagulation for PDR (60) or mild PDR (61) | 7 |
| 65 | Moderate PDR | 8 |
| 71, 75 | High-Risk PDR | 9 |
| 81, 85 | High-Risk PDR with vitreous hemorrhage | 10 |

### **6.2 Sample Size Estimation**

Based on data from eyes with baseline retinopathy in the ACCORD study, it is anticipated that approximately 50% of PROMINENT study participants will have minimal to severe NPDR (levels 20-53) in at least one eye. Among participants with minimal to severe NPDR in at least one eye, the percentage of patients with either a 3-step patient-level progression or photocoagulation was approximately 5% in the fenofibrate group and 12% in the placebo group. For the entire ACCORD cohort (i.e. with and without baseline retinopathy), the rate of DME worsening on color photographs was approximately 3% over 4 years in both the fenofibrate and control groups. However, the percentage of patients with baseline retinopathy and worsening DME without worsening retinopathy is not reported. In addition, DME progression in ACCORD was assessed by color photographs while in the current study it will be assessed by OCT, which has been shown to be more sensitive at detecting DME.<sup>32</sup> Therefore, it is unknown what impact the primary outcome components, besides retinopathy progression, will have on the projected outcome, resulting in uncertainty around these estimates.

The table below shows the required sample size for 80% power with a type I error rate of 5% and a null hypothesis of no difference between groups (two-tailed test) for a time-to-event outcome (log-rank test). These calculations were based on the 4-year outcome rate in the placebo group and the resulting hazard ratio when comparing the outcome rate in the pemafibrate group. The outcome times are assumed to follow an exponential distribution and the estimates include adjustment for 15% attrition over 4 years, also assumed to follow an exponential distribution.

Table 3. Required Number of Participants for Primary Analysis

| Hazard | Placebo Event Rate | | | | |
|--------|--------------------|-----|-----|------|------|
| Ratio | 16% | 14% | 12% | 10% | 8% |
| 0.30 | 270 | 310 | 364 | 438 | 552 |
| 0.40 | 398 | 458 | 536 | 646 | 812 |
| 0.50 | 618 | 710 | 832 | 1000 | 1256 |

The projected 4-year outcome rates of 5% in the pemafibrate group and 12% in the placebo group yield a hazard ratio of approximately 0.4, resulting in a required sample size of 536 participants.

Assuming 600 participants are enrolled of whom 15% are lost to follow up over 4 years, the detectable hazard ratio with 80% power is 0.49 for a placebo event rate of 16% to 0.32 for a placebo event rate of 8%. In other words, the study is powered for a reduction in the rate of diabetic retinopathy worsening by 1/2 to 2/3, depending on the event rate in the placebo group. The placebo event rate could be higher than 16% because the 12% estimate from ACCORD accounts for events due only to progression of retinopathy on photographs and does not include treatment-related and DME-related events, which are other components of the composite outcome. There are no existing data on which to base estimates for rates of these outcomes. In the event that the outcome rates in the placebo group are higher than projected, the study will be powered to detect smaller reductions in the hazard of diabetic retinopathy worsening. Therefore, the estimates given here are conservative.

## 6.3 Primary Analysis Plan

# **6.3.1** Principles for Analysis

The primary treatment group comparison will be based on the hazard ratio from a Cox proportional hazards regression model that adjusts for the baseline person-level retinopathy, which accounts for the retinopathy level in the non-study eye of unilateral participants (see **Table 1**). The primary analysis is an intention-to-treat analysis. Data from participants who are not observed to meet outcome criteria and who are lost to follow up will be censored at the time of the last completed visit. All model assumptions, including proportional hazards, will be verified. If model assumptions are not reasonably satisfied, alternative approaches will be explored.

# 6.3.2 Confounding

Imbalances between groups in important covariates are not expected to be of sufficient magnitude to produce confounding. However, the presence of confounding will be evaluated in regression models by including factors potentially associated with the outcome for which there is an imbalance between groups.

#### **6.3.3** Per Protocol Analyses

Per protocol analyses mimicking the primary intention-to-treat analyses will be performed on the following cohorts:

- Participants with no major protocol deviations as defined by the PROMINENT trial.
- Participants with ≥ 80% compliance during the treatment period as defined by the PROMINENT trial.

#### **6.3.4** Sensitivity Analyses

The following sensitivity analyses will be conducted:

• Repeat the primary analysis while censoring data from participants who receive treatment for DME when the OCT central subfield thickness in the treated eye did not meet the outcome criteria for DME with vision loss when the treatment was given. Participants who do not have an OCT scan from the visit at which treatment is given also will be censored in this analysis.

#### 6.3.5 Subgroup Analyses

The treatment effect in subgroups defined by baseline factors will be assessed in pre-planned subgroup analyses. These analyses will be conducted to determine whether the treatment effect in any subgroup differs from the overall treatment effect. The study is not expected to have sufficient statistical power for definitive conclusions in subgroups and statistical power will be low to formally test for the presence of subgroup effects. Interpretation of subgroup analyses will depend on whether the overall analysis demonstrates a significant treatment effect. In the absence of a significant treatment effect in the primary analysis, assessment of subgroups will be considered exploratory and used to suggest hypotheses for further investigation in future studies.

The general approach for these analyses will be to add an interaction term for the subgroup factor by treatment group into the proportional hazards model used for the primary analysis.

The planned subgroups for analyses are as follows:

• Baseline person-level retinopathy level: Steps 2-4, Steps 5-6, Steps 7-9, and Steps 10-11

Statistical analyses will only be conducted for a subgroup if there are at least 20 participants in each treatment group for that subgroup. The above subgroups are considered those of primary interest for which a rationale for a subgroup effect is hypothesized. The hypothesized mechanism and direction of effect are listed in the table below.

| Factor | Hypothesized direction/mechanism of association |
|---|---|
| Retinopathy Level | Participants with more severe retinopathy have higher risk for |
| | retinopathy worsening and may have disease that is too advanced for the |
| | treatment to work. Therefore, it is possible that the treatment effect is |
| | greater in eyes with less severe disease. |

The following baseline subgroup factors also will be evaluated in exploratory analyses:

- Prior DME treatment: yes vs. no
- Age:  $< 65 \text{ vs.} \ge 65$ 
  - HbA1c: < 7.5% vs.  $\ge 7.5\%$
  - Sex
  - Race/Ethnicity
  - Hyperlipidemia status: ≥ HDL (high-density lipoprotein) median of the sample cohort and ≥ TG (triglyceride) median; ≥ HDL median and < TG median; < HDL median and ≥ TG median; < HDL median and < TG median</li>
  - Number of study eyes: 1 vs. 2

There is no known mechanism supporting an interaction of these effects with treatment group. If a significant subgroup effect for any of these factors is found, it will be interpreted as hypothesis generating only and in need of confirmation from further studies. In particular, there are no data to suggest that the treatment effect will vary by sex or race/ethnicity, although both of these factors will be evaluated.

For all analyses, P-values will be computed for factors based on continuous or ordinal data when available in addition to the categorizations listed above.

#### 6.4 Secondary Outcomes and Safety Outcomes for Treatment Group Comparison

Secondary outcomes will be compared at the 2-year and 4-year visits with the exception of time-to-event outcomes in which the hazard rates will be compared over 4 years only. Safety outcomes collected as part of this ancillary study will be compared at 4 years only. To control for potential correlations arising from participants with two study eyes, eye-level outcomes will be compared using linear mixed models (continuous outcomes), logistic regression using generalized estimating equations (binary outcomes), or Cox proportional hazards regression with a robust sandwich estimate of the covariance matrix (time-to-event outcomes).<sup>33</sup> Participant-level outcomes will be compared similarly but without adjustment for inter-eye correlation.

All analyses will include adjustment for the baseline level of the outcome, where appropriate. In addition, participant-level and eye-level secondary outcomes will be adjusted for baseline person-level diabetic retinopathy severity. The treatment groups will be compared on the following outcomes of interest:

<u>Participant-Level Secondary Outcomes</u> (relates to either eye for bilateral participants and to the study eye for unilateral participants):

- Hazard rate of 3-step person-level (for bilateral participants, **Table 1**) or 2-step eye-level (for unilateral participants, **Table 2**) diabetic retinopathy worsening on the ETDRS Retinopathy Severity Scale or receiving treatment for PDR in at least one study eye at any time (irrespective of DME status or treatment)
  - Percentage of participants with diabetic retinopathy worsening at 2 years and 4 years will be enumerated without statistical comparison
  - Percentage of participants receiving treatment for PDR in at least one study eye at or prior to 2 years and 4 years will be enumerated without statistical comparison
- Hazard rate of developing central-involved DME on OCT with vision loss (as defined in Section 6.1) or receiving treatment for DME in at least one study eye at any time (irrespective of diabetic retinopathy severity level or treatment)
  - Percentage of participants with central-involved DME on OCT with vision loss in at least one study eye at 2 years and 4 years will be enumerated without statistical comparison
  - o Percentage of participants receiving treatment for DME in at least one study eye at or prior to 2 years and 4 years will be enumerated without statistical comparison
- Person-level diabetic retinopathy severity at 2 years and 4 years
- Percentage of participants with at least a 2-line loss in visual acuity from baseline in at least one study eye at 2 years and 4 years

Eye-Level Secondary Outcomes (evaluated only for study eyes):

Hazard rate of a composite PDR/DME outcome. Defined as the time to 2-step diabetic retinopathy worsening on the ETDRS Retinopathy Severity Scale for Individual Eyes (Table 2) at 2 years or 4 years, development of central-involved DME on OCT with vision loss (as defined in Section 6.1) at 2 years or 4 years, or treatment for DME or PDR at any time

 Percentage of eyes with 2-step diabetic retinopathy worsening or development of central-involved DME on OCT with vision loss at 2 years and 4 years will be enumerated without statistical comparison

Safety Outcomes:

- O Percentage of eyes receiving treatment for PDR or DME at or prior to 2 years and 4 years will be enumerated without statistical comparison
- Hazard rate of 2-step diabetic retinopathy worsening or receiving treatment for PDR at any time (irrespective of DME status or treatment)
  - o Percentage of eyes with 2-step diabetic retinopathy worsening at 2 years and 4 years will be enumerated without statistical comparison
  - O Percentage of eyes receiving treatment for PDR at or prior to 2 years and 4 years will be enumerated without statistical comparison
- Hazard rate of developing central-involved DME on OCT with vision loss at 2 years or 4 years or receiving treatment for DME at any time (irrespective of diabetic retinopathy level or treatment)
  - Percentage of eyes with central-involved DME on OCT with vision loss at 2 years and 4 years will be enumerated without statistical comparison
  - o Percentage of eyes receiving treatment for DME at or prior to 2 years and 4 years will be enumerated without statistical comparison
- Eye-level diabetic retinopathy severity at 2 years and 4 years
- Change in OCT central subfield thickness from baseline at 2 years and 4 years
- Change in visual acuity letter score from baseline at 2 years and 4 years
- Percentage of eyes with at least 2-line loss in visual acuity from baseline at 2 years and 4 years
- Adverse events collected as part of this ancillary study including vitreous hemorrhage and retinal detachment
- Changes from randomization in ALT, AST, CK, and creatinine
- To help control the type I error rate at 5%, P-values for secondary outcomes and safety outcomes will be adjusted using the adaptive false discovery rate method of Benjamini and Hochberg in separate sets (i.e., one adjustment for patient-level secondary outcomes, one adjustment for eyelevel secondary outcomes, and one adjustment for safety outcomes).<sup>34</sup> It is recognized that this does not completely control the type I error rate.
- All model assumptions will be verified. These include but are not limited to proportional hazards, linearity, normality of residuals, and homoscedasticity. If model assumptions are not reasonably satisfied, then a transformation of the data or an alternative approach may be considered. Methods for handling missing secondary outcome data will be included in the detailed Statistical Analysis Plan.
- Adverse events reported in this ancillary study as defined in section 4.3 will be enumerated in patient listings and summarized in tables by System Organ Class, using MedDRA terms. Changes in ALT, AST, CK, and creatinine will be depicted as shift tables (i.e., as a shift to high, low, or normal) for each parameter at 4 years.

#### DATA COLLECTION AND MONITORING

### 7.1 Case Report Forms

The key study data are collected through a combination of electronic case report forms (CRFs) and grading of retinal images.

When data are directly collected in electronic case report forms, this will be considered the source data. Each participating site will maintain appropriate medical and research records for this trial, in compliance with ICH E6 and regulatory and institutional requirements for the protection of confidentiality of participants.

#### 7.2 Study Records Retention

Study documents should be retained by the investigator for the latest of 3 years following the end of the current DRCR.net grant, 2 years after the last approval of a marketing application, and until there are no pending or contemplated marketing applications, or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents should be retained for a longer period, however, if required by local regulations. No records will be destroyed without the written consent of the Jaeb Center for Health Research. It is the responsibility of the sponsor to inform the investigator when these documents no longer need to be retained.

### 7.3 Quality Assurance and Monitoring

Designated personnel from the JCHR Coordinating Center will be responsible for maintaining quality assurance and quality control systems to ensure that the clinical portion of the trial is conducted and data are generated, documented and reported in compliance with the protocol, Good Clinical Practice (GCP) and the applicable regulatory requirements.

A risk-based monitoring plan will be developed and revised as needed during the course of the study, consistent with the FDA "Guidance for Industry Oversight of Clinical Investigations — A Risk-Based Approach to Monitoring" (August 2013).

The data of most importance for monitoring at the site are participant eligibility and image outcome data. Therefore, the risk-based monitoring plan will focus on these areas. As much as possible, remote monitoring will be performed in real-time with on-site monitoring performed to evaluate the verity and completeness of the key site data when possible. Elements of the risk-based monitoring will include:

- Qualification assessment, training, and certification for sites and site personnel
- Oversight of Institutional Review Board (IRB) coverage and informed consent procedures
- Central (remote) data monitoring: validation of data entry, data edits/audit trail, protocol review of entered data and edits, statistical monitoring, study closeout
- On-site monitoring (site visits): source data verification, site visit report
- Communications with site staff
- Patient retention and visit completion
- Quality control reports
- Management of noncompliance
- Documenting monitoring activities
- Adverse event reporting and monitoring

JCHR Coordinating Center representatives or their designees may visit the study facilities at any time in order to maintain current and personal knowledge of the study through review of the records, comparison with source documents, observation and discussion of the conduct and progress of the study.

850 851

852

853

854

#### 7.4 Protocol Deviations

A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or procedure requirements. The noncompliance may be either on the part of the participant, the investigator, or the study site staff. As a result of deviations, corrective actions are to be developed by the site and implemented promptly.

855856857

858859

The site principal investigator/study staff is responsible for knowing and adhering to their IRB requirements. Further details about the handling of protocol deviations will be included in the monitoring plan.

#### ETHICS/PROTECTION OF HUMAN PARTICIPANTS

#### 8.1 Ethical Standard

The investigator will ensure that this study is conducted in full conformity with Regulations for the Protection of Human Participants of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, and/or the ICH E6.

#### 8.2 Institutional Review Boards

The protocol, informed consent form, recruitment materials, and all participant materials will be submitted to the IRB for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. All changes to the consent form will be IRB approved; a determination will be made regarding whether previously consented participants need to be re-consented.

#### **8.3 Informed Consent Process**

#### **8.3.1** Consent Procedures and Documentation

Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study and continues throughout the individual's study participation. Extensive discussion of risks and possible benefits of participation will be provided to the participants and their families. Consent forms will be IRB-approved and the participant will be asked to read and review the document. The investigator will explain the research study to the participant and answer any questions that may arise. All participants will receive a verbal explanation in terms suited to their

questions that may arise. All participants will receive a verbal explanation in terms suited to their comprehension of the purposes, procedures, and potential risks of the study and of their rights as

research participants. Participants will have the opportunity to carefully review the written consent

form and ask questions prior to signing.

The participants should have the opportunity to discuss the study with their surrogates or think about it prior to agreeing to participate. The participant will sign the informed consent document prior to any procedures being done specifically for the study. The participants may withdraw consent at any time throughout the course of the trial. A copy of the informed consent document will be given to the participants for their records. The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

# 8.3.2 Participant and Data Confidentiality

Participant confidentiality is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their agents. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence.

The study monitor, other authorized representatives of the sponsor or, representatives of the IRB may inspect all documents and records required to be maintained by the investigator, including but not limited to medical records (office, clinic, or hospital). The clinical study site will permit access to such records.

The study participant's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure

location for as long a period as dictated by local IRB and Institutional regulations.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the JCHR Coordinating Center. This will not include a link to

907 the participant's contact or identifying information. Rather, individual participants and their

research data will be identified by a unique study identification number. The study data entry and

- study management systems used by clinical sites and by JCHR Coordinating Center research staff will be secured and password protected. At the end of the study, all study databases will be deidentified and archived at the JCHR Coordinating Center. 909 910
- 911

#### REFERENCES

- 1. Centers for Disease Control and Prevention. State-specific incidence of diabetes among adults--participating states, 1995-1997 and 2005-2007. *MMWR Morb Mortal Wkly Rep.* 2008;57(43):1169-73.
- 2. International Diabetes Federation: Facts and figures. <a href="http://www.idf.org/worlddiabetesday/toolkit/gp/facts-figures">http://www.idf.org/worlddiabetesday/toolkit/gp/facts-figures</a> Accessed 26 September 2016.
- 3. Vision problems in the U.S.: Prevalence of adult vision impairment and age-related eye disease in America. http://www.visionproblemsus.org/. Accessed 16 November 2016.
- **4.** Antonetti DA, Klein R, Gardner TW. Diabetic retinopathy. *N Engl J Med.* 2012;366(13):1227-39.
- **5.** Aiello LP. Angiogenic pathways in diabetic retinopathy. *N Engl J Med.* 2005;353:839-41.
- 6. Davis MD, Fisher MR, Gangnon RE, et al. Risk factors for high-risk proliferative diabetic retinopathy and severe visual loss: Early Treatment Diabetic Retinopathy Study Report #18. *Invest Ophthalmol Vis Sci.* 1998;39(2):233-52.
- 7. Stratton IM, Kohner EM, Aldington SJ, et al. UKPDS 50: risk factors for incidence and progression of retinopathy in Type II diabetes over 6 years from diagnosis. *Diabetologia*. 2001;44(2):156-63.
- **8.** Chew EY, Ambrosius WT, Davis MD, et al. Effects of medical therapies on retinopathy progression in type 2 diabetes. *N Engl J Med.* 2010;363(3):233-44.
- 9. The Diabetes Control and Complication Trial Research Group. The effect of intensive treatment of diabetes on the development and progression of long-term complication in insulin-dependent diabetes mellitus. *N Engl J Med.* 1993;329:977-86.
- 10. The Diabetes Control and Complication Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Retinopathy and nephropathy in patients with type 1 diabetes four years after a trial of intensive therapy. The Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. *N Engl J Med.* 2000;342(6):381-9.
- 11. Diabetes Control Complications Trial /Epidemiology of Diabetes Interventions Complications Research Group, Lachin JM, White NH, et al. Effect of intensive diabetes therapy on the progression of diabetic retinopathy in patients with type 1 diabetes: 18 years of follow-up in the DCCT/EDIC. *Diabetes*. 2015;64(2):631-42.
- **12.** Dcct Edic Research Group, Aiello LP, Sun W, et al. Intensive diabetes therapy and ocular surgery in type 1 diabetes. *N Engl J Med.* 2015;372(18):1722-33.
- **13.** Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. *N Engl J Med.* 2008;359(15):1577-89.
- 14. Action to Control Cardiovascular Risk in Diabetes Follow-On Eye Study G, the Action to Control Cardiovascular Risk in Diabetes Follow-On Study G. Persistent Effects of Intensive Glycemic Control on Retinopathy in Type 2 Diabetes in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Follow-On Study. *Diabetes Care*. 2016;39(7):1089-100.
- 15. Klein R, Klein BE. Are individuals with diabetes seeing better?: a long-term epidemiological perspective. *Diabetes*. 2010;59(8):1853-60.
- **16.** Centers for Disease Control and Prevention. National Diabetes Fact Sheet. <a href="https://www.cdc.gov/visionhealth/pdf/factsheet.pdf">https://www.cdc.gov/visionhealth/pdf/factsheet.pdf</a>, Accessed March 21, 2011.
- 17. Avery RL, Pearlman J, Pieramici DJ, et al. Intravitreal bevacizumab (Avastin) in the treatment of proliferative diabetic retinopathy. *Ophthalmology*. 2006;113(10):1695 e1-15.
- **18.** Diabetic Retinopathy Clinical Research Network. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. *Ophthalmology*. 2010;117(6):1064-77 e35.

- 19. Writing Committee for the Diabetic Retinopathy Clinical Research Network, Gross JG, Glassman AR, et al. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. *JAMA*. 2015;314(20):2137-46.
- **20.** Sampat KM, Garg SJ. Complications of intravitreal injections. *Curr Opin Ophthalmol*. 2010;21(3):178-83.
- **21.** Diabetic Retinopathy Clinical Research Network, Wells JA, Glassman AR, et al. Aflibercept, bevacizumab, or ranibizumab for diabetic macular edema. *N Engl J Med*. 2015;372(13):1193-203.
- **22.** American Academy of Ophthalmology. *Preferred practice pattern diabetic retinopathy*. San Francisco: American Academy of Ophthalmology; 1998.
- **23.** Hiukka A, Maranghi M, Matikainen N, Taskinen MR. PPARalpha: an emerging therapeutic target in diabetic microvascular damage. *Nat Rev Endocrinol*. 2010;6(8):454-63.
- 24. Noonan JE, Jenkins AJ, Ma JX, Keech AC, Wang JJ, Lamoureux EL. An update on the molecular actions of fenofibrate and its clinical effects on diabetic retinopathy and other microvascular end points in patients with diabetes. *Diabetes*. 2013;62(12):3968-75.
- **25.** Ding L, Cheng R, Hu Y, et al. Peroxisome proliferator-activated receptor alpha protects capillary pericytes in the retina. *Am J Pathol.* 2014;184(10):2709-20.
- **26.** Roy S, Kim D, Hernandez C, Simo R, Roy S. Beneficial effects of fenofibric acid on overexpression of extracellular matrix components, COX-2, and impairment of endothelial permeability associated with diabetic retinopathy. *Exp Eye Res.* 2015;140:124-9.
- 27. Zhao S, Li J, Wang N, et al. Feno fi brate suppresses cellular metabolic memory of high glucose in diabetic retinopathy via a sirtuin 1-dependent signalling pathway. *Mol Med Rep.* 2015;12(4):6112-8.
- **28.** Gong Y, Shao Z, Fu Z, et al. Fenofibrate Inhibits Cytochrome P450 Epoxygenase 2C Activity to Suppress Pathological Ocular Angiogenesis. *EBioMedicine*. 2016;13:201-11.
- **29.** Farris RA, Price ET. Reverse Translational Study of Fenofibrate's Observed Effects in Diabetes-Associated Retinopathy. *Clin Transl Sci.* 2017;10(2):110-6.
- **30.** Keech AC, Mitchell P, Summanen PA, et al. Effect of fenofibrate on the need for laser treatment for diabetic retinopathy (FIELD study): a randomised controlled trial. *Lancet*. 2007;370(9600):1687-97.
- 31. Chew EY, Davis MD, Danis RP, et al. The effects of medical management on the progression of diabetic retinopathy in persons with type 2 diabetes: the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Eye Study. *Ophthalmology*. 2014;121(12):2443-51.
- **32.** Davis MD, Bressler SB, Aiello LP, et al. Comparison of time-domain OCT and fundus photographic assessments of retinal thickening in eyes with diabetic macular edema. *Invest Ophthalmol Vis Sci.* 2008;49(5):1745-52.
- 33. Lee EW, Wei LJ, Amato DA. *Cox-type regression analysis for large numbers of small groups of correlated failure time observations*: Dordrecht: Kluwer Academic; 1992.
- 34. Benjamini Y, Hochberg Y. On the Adaptive Control of the False Discovery Rate in Multiple Testing With Independent Statistics. *Journal of Educational and Behavioral Statistics*. 2000;25(1):60-83.